CLINICAL TRIAL: NCT01687049
Title: A Prospective Study of Red Yeast Rice in Subjects With Clinically Localized Prostate Cancer Undergoing Active Surveillance
Brief Title: Red Yeast Rice in Subjects With Clinically Localized Prostate Cancer Undergoing Active Surveillance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Laurence Klotz (Other)
Responsible Party: Sponsor-Investigator, Dr. Laurence Klotz, Principal Investigator, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REALITY; SHSC (Other: Urology Research, Sunnybrook Health Sciences Centre)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Prostate Cancer
Keywords: nonmetastatic; localized; prostate; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — red yeast rice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- red yeast rice (RYR) (Experimental): Two RYR capsules three times daily for a minimum of 6 months
  Interventions: Drug: Red yeast rice

INTERVENTIONS:
Drug: Red yeast rice
  Other Names: Aliperol

SUMMARY:
Agents that inhibit cholesterol synthesis are being investigated in cancers dependent upon cholesterogenesis. Red yeast rice (RYR), is a reddish-purple fermented rice, containing statins which are known to inhibit cholesterol synthesis. Laboratory studies have also shown that RYR has direct effects on androgen dependent and androgen independent prostate cancer cells, inhibiting their growth. It is thought that RYR may have clinical benefit in those subjects with localized prostate cancer who have chosen to be managed by active surveillance.

DETAILED DESCRIPTION:
Red yeast rice has been promoted as a safe and effective alternative to statin therapy in the treatment of hypercholesterolemia. Red yeast rice has the potential to slow prostate cancer growth by inhibiting cholesterol and androgen biosynthesis. There is a strong rationale for the use of RYR in patients being managed with active surveillance for localized, low risk, prostate cancer. To date, no human studies utilizing RYR in this setting have been reported.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosis of prostate adenocarcinoma
* being monitored by active surveillance for favourable risk prostate cancer
* tumour material from most recent prostate biopsy available with sample
* scheduled to have an active surveillance mandated transrectal ultrasound (TRUS) guided biopsy within 6 - 12 months of Day 1 of the study

Exclusion Criteria:

* previous malignancy in the past 5 years
* no previous or concurrent treatment for prostate cancer
* inability to undergo TRUS biopsy
* ECOG > 2
* known or previous history of liver disease

Ages: 19 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Expression of Ki-67 and p27 biomarkers | 6 months
  Determine effect of red yeast rice therapy on expression of ki67 and p27 biomarkers in a post-treatment biopsy

SECONDARY OUTCOMES:
PSA kinetics | 6 months
  Determine effect of red yeast rice daily therapy on PSA kinetics in men on active surveillance for localized prostate cancer
Presence of prostatic interepithelial neoplasia | 6 months
  To evaluate the effect of red yeast rice daily therapy on grade and the presence of prostatic intraepithelial neoplasia (PIN) in post treatment biopsy
Expression of hs-CRP and cardiac CRP | 6 months
  To assess the effect of red yeast rice therapy on the expression of high sensitivity C-reactive protein (hs-CRP) and cardiac C-reactive protein (CRP) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada